CLINICAL TRIAL: NCT06224556
Title: A Personalized Prevention Program (PPP) Based on the Comprehensive Geriatric Assessment (CGA) for the Prevention of Multidimensional Frailty Related to Non-communicable Chronic Diseases (NCDs) in Older People: a Practical Approach in Primary Care Setting
Brief Title: A Personalized Prevention Program (PPP) Based on the Comprehensive Geriatric Assessment (CGA) for the Prevention of Multidimensional Frailty Related to Non-communicable Chronic Diseases (NCDs) in Older People
Acronym: PrimaCare_P3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alberto Pilotto (Other)
Responsible Party: Sponsor-Investigator, Alberto Pilotto, Director of Department of Geriatric Care, Orthogeriatrics and Rehabilitation, Ente Ospedaliero Ospedali Galliera
Organization: Ente Ospedaliero Ospedali Galliera (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PNRR-MAD-2022-12376781
Record Dates: First submitted 2024-01-05; First posted 2024-01-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Older People; Non-Communicable Chronic Diseases
Keywords: Primary care setting; Comprehensive Geriatric Assessment; Older people; Non-communicable chronic diseases; Personalized Prevention Program; Saliva collection
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: The Intervention Group will receive the Personlized Prevention Program (PPP)
  be evaluated by a Comprehensive Geriatric Assessment thanks to the Multidimensional Prognostic Index (MPI) questionnaire.
Who Masked: Care Provider
Masking Description: The General Practitioners (GPs) involved will be randomised in clusters in a 1:1 ratio, therefore one group of GPs will enrol patients for the Intervention Group and a second group of GPs will include patients for the Control Group.
  Therefore, the role of GPs are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): All the 608 patients will be evaluated by their General Practitioners through the Brief-MPI scale, which is based on the Comprehensive Geriatric Assessment (CGA).
  Based on the score obtained at the Brief-MPI, the patient will receive a Personalised Prevention Program (PPP) concerning the following domains: 1) motor, 2) cognitive, 3) nutritional, 4) polypharmacotherapy, 5) vaccination prevention, 6) basal and instrumental activities, 7) co-habitation. Patients will receive brochures containing practical advice and recommendations to be implemented over a 12-month period; in the case of high Brief-MPI risk scores, patients will be referred for specialist examinations and/or in-depth diagnostics.
  In addition, saliva samples will be collected to assess biomarkers of oxidative stress and, in a subsample of 210 subjects, the composition of the oral microbiota will also be analysed.
  Interventions: Combination Product: Brief-MPI assessment (based on the Comprehensive Geriatric Assessment); Personalized Prevention Program
- Control group (No Intervention): Patients will receive the standard clinical practice by their General Practitioners, without being evaluated by the CGA or receiving the personalized prevention program (PPP). No saliva sample will be collected.

INTERVENTIONS:
Combination Product: Brief-MPI assessment (based on the Comprehensive Geriatric Assessment); Personalized Prevention Program — Patients will be evaluated at baseline and at 6 and 12 months after the baseline through the CGA, the Resilience Scale (RS-14 items) and the Psychological General Wellbeing Index short form.
  The prevention program will be received at the baseline, so at the two follow-ups patients wiil asked the adherence to it and the level of satisfaction (Client Satisfaction Questionnaire - 8 items).
  Saliva sample will be collected and analyzed.
  Arms: Intervention Group

SUMMARY:
* Non-Communicable Diseases (NCDs) can accelerated the aging process and increase the frailty condition
* The Comprehensive Geriatric Assessment (CGA) is the gold standard in the geriatric clinical context
* Recently, in Italy the first Guidelines about the CGA in different settings for older people has been pubblicated
* The CGA can identify older people at high risk of frailty who can benefit from a personalized prevention program
* No studies has been investigated the effects of a personalized prevention program (PPP) based on the CGA in a primary care setting
* The main hypothesis is that the CGA assessment can result in personalized prevention programs for older subjects in primary care settings with an effect in reducing the hospitalization rate and can be related to the biological paramters in NCDs

DETAILED DESCRIPTION:
The main aim of the project is to evaluate in older people the effectiveness of personalized preventive interventions based on the Comprehensive Geriatric Assessment (CGA) in the primary care setting and to explore biological process in Non-Communicable Disases (NCDs).

The study involves 1216 subjects enrolled by General Practitioners (GPs) in four different Italian Areas.

The GPs involved will be randomised to clusters in a 1:1 ratio, therefore one group of GPs will enrol patients for the Intervention Group and a second group of GPs will include patients for the Control Group.

The sample size:

A recent Cochrane systematic review reports a significant reduction in the risk of unplanned hospitalisation in community-dwelling elderly persons treated with VMD compared to standard clinical practice (RR= 0.83; CI 95%: 0.70-0.99). Thus, assuming an incidence of unplanned hospitalisations in one year of 38.8% in the group receiving PPP compared to 47.7% in the group randomised to standard care and assuming a power of 80% and a type I error of 5%, a total of 972 participants will be enrolled. Furthermore, assuming a drop-out rate of 20% over the 1-year follow-up period, the final sample will be 1216 participants, 608 in each group

608 subjects will be involved in the intervention group: they will receive the Personalized Prevention Program (PPP) and a saliva sample will be collected.

608 subjects will be involved in the control group according to the normal clinical practice.

Both groups will be contacted at 6 and 12 months after the baseline for the follow-up.

Statistical analyses:

Baseline characteristics will be compared between the group receiving the CGA-based PPP intervention and the control group. Continuous variables will be compared using the t-Student test and categorical variables using the Chi-square test. The cumulative probability of the primary and secondary outcome will be estimated by Kaplan-Meier curve, using the log-rank test to assess differences between the two groups. To assess the risk associated with the primary outcome (rate of unplanned hospitalisation at 12 months) in subjects in the intervention group compared to subjects in standard care, the Hazard Ratio (HR) will be estimated by fitting a Cox model, after testing for proportional hazards. Similarly, the risk of secondary outcomes will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old and over
* At least 1 non-communicable chronic disease
* Signed informed consent

Exclusion Criteria:

* not willing in partecipating in the study and no signed informed consent
* <65 years old
* without non-communicable chronic diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1216 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate | 12 months
  Unplanned hospitalization rate

SECONDARY OUTCOMES:
Composed outcome | 6 and 12 months
  Composed outcome including: emergency access rate, hospitalization and institutionalization rates at 6 and 12 months after the baseline.
Number of unplanned General Practitioners visits | 12 months
  Unplanned GPs visits
Mortality rate | 6 and 12 months
  mortality rate at 6 and 12 months

OTHER OUTCOMES:
Adherence at the PPP | 6 and 12 months
  Adherence at the Personalized Prevention Program by the Intervention Group
Psychological Well-being | Baseline, 6 and 12 months
  Psychological well-being assessed to the Intervention Group
Resilience | Baseline, 6 and 12 months
  Resilience outcome evaluated in the Intervention Group
Lactate in the Intervention Group | After the saliva collection at the baseline
  Saliva analyses for the Lactate parameter
NAD/NADH in the Intervention Group | After the saliva collection at the baseline
  Saliva analyses for theNAD/NADH parameter
TBARS in the Intervention Group | After the saliva collection at the baseline
  Saliva analyses for the TBARS parameter
TNF-alfa in the Intervention Group | After the saliva collection at the baseline
  Saliva analyses for theTNF-alfa parameter
IL-1b in the Intervention Group | After the saliva collection at the baseline
  Saliva analyses for the IL-1b parameter
IL-6 in the Intervention Group | After the saliva collection at the baseline
  Saliva analyses for the IL-6 parameter
IL-8 in the Intervention Group | After the saliva collection at the baseline
  Saliva analyses for the IL-8 parameter
Microbioma saliva analysis in a sub-group of the Intervention Group | After the saliva collection at the baseline
  The microbioma saliva sample will be analysed in 210 subjects from the Intervention Group through the DNA GENOTEK OME-505 Omnigene Oral Collection Kits for Nucleic Acid Saliva

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pilotto, Principal Investigator — Director of the Department of Geriatric Care, orthogeroatric and rehabilitation, EO Galliera Hospital, Genova, Italy
Locations (4):
- Italy (4):
  - Polimedica Societa' Cooperativa, Bari
  - Medici Insieme Garda Valsabbia Societa' Cooperativa, Desenzano del Garda
  - Ambulatori medici, Florence
  - COMEGEN Società Cooperativa Sociale, Napoli

IPD SHARING:
Plan to Share IPD: No
Results referred to the groups of subjects will be published in one or more different papers with only statistically significant data with the description of statistical methods of the analyses. No individual or personal data will be shared.

REFERENCES:
- [Derived] Pilotto A, Morganti W, Seminerio E, Lacorte E, Custodero C, Veronese N, Fielding P, Massone C, Piscopo P, Fabrizi E, Lorenzini P, Magni A, Piccinocchi G, Ignazzi C, Busco L, Barbagallo M, Massone C, Aprile PL, Vanacore N. Usefulness of the BRIEF-Multidimensional Prognostic Index (BRIEF-MPI) to identify older adults' healthcare needs to be addressed with a Personalized Prevention Program in general practice: preliminary data from the PrimaCare_P3 study. BMC Prim Care. 2025 Oct 27;26(1):323. doi: 10.1186/s12875-025-02951-6. PMID 41146026
- [Derived] Pilotto A, Barbagelata M, Lacorte E, Custodero C, Veronese N, Maione V, Morganti W, Seminerio E, Piscopo P, Fabrizi E, Lorenzini P, Carbone E, Lora Aprile P, Solfrizzi V, Barbagallo M, Vanacore N; PrimaCare_P3 study group. A multicomponent personalized prevention program in the primary care setting: a randomized clinical trial in older people with noncommunicable chronic diseases (Primacare_P3 study). Trials. 2024 Sep 13;25(1):611. doi: 10.1186/s13063-024-08413-1. PMID 39272196